CLINICAL TRIAL: NCT06675500
Title: Evaluation of the Role of Magnesium in Prevention of AF Post Cardiac Surgery
Acronym: Magnesium AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, sarah hamdy, lecturer of Anesthesia, Intensive Care and Pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU R255/2024
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Results first posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Atrial Fibrillation (AF); Magnesium Sulfate; Post Cardiac Surgery Patients
Keywords: magnesium sulphate; post cardiac surgery arrhythmia; atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: This study is a prospective, randomized controlled trial that will study the postoperative anti-arrhythmic effect of Magnesium Sulfate and clinical outcomes of administration of intravenous Mg Sulfate in patients undergoing open heart surgery.
  Randomization will be performed using a computer-generated randomization sequence and allocation concealment to be maintained all through the time of procedure, by using opaque, numbered, and sealed envelopes.
  Informed consent will be obtained from each patient before patients' allocation.
  Patients will be randomly allocated by computer generated randomization into two groups A and B.
  After completion of surgical procedure and successful weaning off Cardiopulmonary bypass the patients will be divided into two groups group A will receive 2 gm of Mg Sulfate diluted in 30 cc normal 0.9 % saline via intravenous infusion over 1 hour (1 Mg sulfate ampoule = 10 cc) and group B will receive 50 cc normal 0.9 % saline via intravenous infusion.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Study group) (Active Comparator): After completion of surgical procedure and successful weaning off Cardiopulmonary bypass the patients will be divided into two groups group A will receive 2 gm of Mg Sulfate diluted in 30 cc normal 0.9 % saline via intravenous infusion over 1 hour (1 Mg sulfate ampoule = 10 cc) .
  On ICU arrival group A will continue receiving 1 gm of Mg sulfate per hour for five hours via continuous IV infusion.
  After 5 hours, group A will receive 200 mg of Mg sulfate per hour for 19 hours via continuous IV infusion, then oral replacement of mag added 1 gm/8 hours tablet.
  Total time of Mg/placebo infusion is 24 hours, and oral tablets for 1 week just before hospital discharge.
  Total serum Magnesium level will be measured immediately post weaning of cardiopulmonary bypass, on ICU arrival, after 24 and 48 hours.
  Interventions: Drug: Magnesium sulphate
- Group B (Control group) (Placebo Comparator): After completion of surgical procedure and successful weaning off Cardiopulmonary bypass the patients will be divided into two groups group B will receive 50 cc normal 0.9 % saline via intravenous infusion over same period.
  On ICU arrival group B will same volume and rate of normal saline. After 5 hours, group B will receive same fluid volume and rate of normal saline followed by oral inert starch tablets.
  Total time of Mg/placebo infusion is 24 hours, and oral tablets for 1 week just before hospital discharge.
  Total serum Magnesium level will be measured immediately post weaning of cardiopulmonary bypass, on ICU arrival, after 24 and 48 hours.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Magnesium sulphate — Intravenous Magnesium sulphate followed by oral tablets of Magnesium sulphate
  Arms: Group A (Study group)
Drug: Placebo — Intravenous infusion of Normal saline 0.9 followed by starch oral tablets
  Arms: Group B (Control group)

SUMMARY:
Atrial fibrillation (AF) is a common complication after cardiac surgery. Most studies suggest that the frequency ranges between 25-40%.

Some studies have shown that serum hypomagnesaemia is common after coronary artery bypass grafts (CABG) and other types of cardiac surgery and is associated with postoperative morbidity such as atrial tachyarrhythmia.

The aim of the present study is to investigate the anti-arrhythmic effect of Magnesium Sulfate in prevention of atrial fibrillation post cardiac surgery.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is a common complication after cardiac surgery. Most studies suggest that the frequency ranges between 25-40%.

Several reports have indicated that postoperative AF is associated with an increased length of in-hospital stay (LOS) and consequently a greater utilization of health care resources.

Postoperative AF is also associated with higher rates of postoperative stroke, compromised cardiac function, and adverse effects from drugs used to prevent AF.

Despite many years of clinical experience and a large amount of investigation, prevention, and treatment of postoperative AF remain controversial. Many questions about the mechanisms and pathophysiology of AF remain unanswered, further contributing to the ambiguity in reaching consensus about appropriate treatment. Increasing patient age, valvular lesion and dilated atrial diameter is generally considered the greatest risk factor for postoperative AF and an aging population suggest that postoperative AF will continue to be a considerable problem in the future.

Magnesium (Mg) is an important intracellular ion with electrophysiological properties. It is essential for optimal metabolic cell function. Mg has proven effective for treating eclampsia, preeclampsia, and torsade's de pointes. Other therapeutic applications such as adjunctive therapy in acute asthma exacerbations, acute coronary syndromes, acute cerebral ischemia, and postoperative pain control are under discussion.

Some studies have shown that serum hypomagnesaemia is common after coronary artery bypass grafts (CABG) and other types of cardiac surgery. and is associated with postoperative morbidity such as atrial tachyarrhythmia.

Some clinical trials have assessed the efficacy of magnesium as a method of intervention to reduce the incidence of postoperative AF. Though this study is a negative one, other studies showed that magnesium sulfate has a body of evidence supporting its anti-arrhythmic effects and safety profile in AF prevention post-surgery.

A Phase III trial is necessary to further validate the efficacy and safety of magnesium sulfate because the previous studies, while promising, have shown varying results and may have methodological limitations such as small sample sizes, lack of rigorous randomization, or not accounting for long-term outcomes. This study aims to provide definitive evidence through a well-powered randomized controlled trial, using more rigorous study designs, thereby filling an important gap in clinical evidence.

The currently considered standard preventive care for AF after cardiac surgery includes the use of beta-blockers, amiodarone, or other antiarrhythmic drugs. These measures can then be contrasted with the magnesium sulfate intervention, highlighting its potential advantages and rationale for testing in this study.

A placebo group is used in this study since magnesium sulfate has shown some benefit in previous studies, the evidence is not definitive. Therefore, a placebo group is necessary to ensure that any observed effects of magnesium sulfate are due to the treatment and not other confounding factors.

ELIGIBILITY:
Inclusion Criteria:

* • Elective open heart surgeries for coronary bypass grafting CABG,valvular lesion single or multiple replacement, combined CABG and valvular; with EF in preoperative echo is more than or equal 40%

Exclusion Criteria:

* Patients refuse to give informed consent.
* Emergency open heart surgeries
* Redo cases.
* Patients with preoperative serum creatinine level ≥ 1.8 mg/dL
* Patients with reduced intra/post operative urine output ≤ 1 ml/kg/hour.
* Patients with Chronic Kidney disease, Renal failure on dialysis
* Patients with rhythm defects as proved by ECG before administration of Mg/Placebo.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine ,Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Miller S, Crystal E, Garfinkle M, Lau C, Lashevsky I, Connolly SJ. Effects of magnesium on atrial fibrillation after cardiac surgery: a meta-analysis. Heart. 2005 May;91(5):618-23. doi: 10.1136/hrt.2004.033811. PMID 15831645
- [Background] Hogue CW Jr, Hyder ML. Atrial fibrillation after cardiac operation: risks, mechanisms, and treatment. Ann Thorac Surg. 2000 Jan;69(1):300-6. doi: 10.1016/s0003-4975(99)01267-9. PMID 10654548
- [Background] Fuller JA, Adams GG, Buxton B. Atrial fibrillation after coronary artery bypass grafting. Is it a disorder of the elderly? J Thorac Cardiovasc Surg. 1989 Jun;97(6):821-5. PMID 2566713

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group A (Study Group) | Group B (Control Group)
Started | 65 | 65
Completed | 65 | 65
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A (Study Group) | Group B (Control Group) | Total
Number analyzed (Participants) | 65 | 65 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.1 (10.3) | 59.0 (9.7) | 58.6 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 37
  Male | 45 | 48 | 93
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With New Episodes of Atrial Fibrillation
Description: Count of participants developing atrial fibrillation (AF) (episode >30 seconds) confirmed by 12-lead ECG or continuous telemetry during hospitalization (≤7 days).
Time Frame: 7 days
Measure: Number; unit: participants
Arm/Group | Group A (Study Group) | Group B (Control Group)
Number analyzed (Participants) | 65 | 65
participants | 12 | 27

2. Secondary Outcome: Total ICU Length of Stay
Description: Total duration of ICU admission from postoperative transfer to discharge, measured in days
Time Frame: From ICU admission until discharge (assessed up to 30 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group A (Study Group) | Group B (Control Group)
Number analyzed (Participants) | 65 | 65
days | 2.1 (0.8) | 3.5 (1.2)

3. Secondary Outcome: Total Ventilation Time
Description: mechanical ventilatory support in hours
Time Frame: 48 hours
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Group A (Study Group) | Group B (Control Group)
Number analyzed (Participants) | 65 | 65
hours | 8.4 (3.1) | 7.8 (2.1)

4. Secondary Outcome: Number of Participants With New Postoperative Renal Impairment
Description: Count of participants meeting ≥1 criterion:
  1. Postoperative serum creatinine ≥1.8 mg/dL
  2. Requirement of renal replacement therapy (hemodialysis, transient, or permanent)
Time Frame: 30 days
Measure: Number; unit: participants
Arm/Group | Group A (Study Group) | Group B (Control Group)
Number analyzed (Participants) | 65 | 65
participants | 4 | 9

ADVERSE EVENTS:
Time Frame: From surgery until hospital discharge, up to 30 days
Description: Adverse events were systematically assessed from surgery until hospital discharge (up to 30 days) using clinical exams, lab tests (creatinine, electrolytes), telemetry, and intervention records. Events were coded using MedDRA v26.0. Note: All participants were monitored for adverse events.
Arm/Group | Group A (Study Group) | Group B (Control Group)
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/65
Serious Adverse Events (participants affected / at risk) | 10/65 | 20/65
Other Adverse Events (participants affected / at risk) | 8/65 | 10/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (Study Group) (N=65) | Group B (Control Group) (N=65)
Renal impairment (Renal and urinary disorders) | 4 | 9
Stroke (Nervous system disorders) | 1 | 2
Reoperation for bleeding (Surgical and medical procedures) | 5 | 9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (Study Group) (N=65) | Group B (Control Group) (N=65)
Hypotension (Cardiac disorders) | 8 (65) | 10 (65)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-11-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT06675500/Prot_SAP_000.pdf